CLINICAL TRIAL: NCT02025361
Title: Impact of Local Anesthesia Type on Cancer Detection Rate in Transrectal Ultrasound Guided Prostate Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Zafer Temiz, principal investigator, Bagcilar Training and Research Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: Cancer detection in TRUS-Bx
Record Dates: First submitted 2013-12-17; First posted 2014-01-01 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Adenocarcinoma of Prostate
Keywords: prostate biopsy, local anesthesia, cancer detection rate.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrarectal lidocaine gel (Experimental): transrectal ultrasound guided prostate biopsy was performed with intrarectal lidocaine gel anesthesia: 10 minutes before the procedure % 2 lidocaine hydrochloride gel instilated into the rectum for local anesthesia
  Interventions: Drug: intrarectal lidocaine gel
- periprostatic nerve blockade (Experimental): transrectal ultrasound guided prostate biopsy was performed with intrarectal lidocaine gel anesthesia: 10 minutes before the procedure transrectal ultrasound guided 10 ml prilocaine and serum physiologic blend (5ml %2 prilocaine and 5 ml serum physiologic) injected separetly 5ml right and 5ml left junction between the prostate base and seminal vesicle.
  Interventions: Drug: periprostatic nerve blockade

INTERVENTIONS:
Drug: intrarectal lidocaine gel — intrarectal local anesthetic application
  Other Names: No name
  Arms: intrarectal lidocaine gel
Drug: periprostatic nerve blockade — periprostatic local anesthetic application
  Other Names: No name
  Arms: periprostatic nerve blockade

SUMMARY:
Transrectal ultrasound guided prostate biopsy (TRUS-Bx) is the gold standard method for prostat cancer diagnosis. Cancer detection rate is an important issue in TRUS-Bx. Effective biopsy protocol is necessary to enhance cancer detection rate during the procedure. Patient tolerance may improve the protocol effectiveness and quality.

Adequate patient tolerance with optimal local anesthesia may enhance cancer detection rate in TRUS-Bx.

DETAILED DESCRIPTION:
In transrectal ultrasound guided prostate biopsy ultrasound's probe manipulation is necessary for effective biopsy. Patient discomfort and pain frequently occurs with manipulation of probe during transrectal ultrasound guided prostate biopsy and this situation may qualify of the achievement of this procedure.

In this study, we aimed to describe the impact of different two local anesthesia types on cancer detection rate in transrectal ultrasound guided prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent transrectal ultrasound guided prostate biopsy because of elevated serum PSA levels and/or suspicious rectal examination of prostate.

Exclusion Criteria:

* Previous TRUS-Bx and prostatic operations(TUR-P, open prostatectomy, etc..) history, treatment for prostate carcinoma, usage of finasteride and dutasteride.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
cancer detection rate with anesthesia type | finally pathologic evaluation within 2-3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: mustafa z temiz, Principal Investigator — bagcilar training and research hospital-depertmant of urology
Locations (1):
- Bagcilar Training and Research Hospital-Depertmant of urology, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No